CLINICAL TRIAL: NCT02992418
Title: Immunogenicity and Safety of a Tetravalent Dengue Vaccine Administered Concomitantly or Sequentially With Adacel® in Healthy Subjects Aged 9 to 60 Years in the Philippines
Brief Title: Study of a Tetravalent Dengue Vaccine Administered Concomitantly or Sequentially With Adacel® in Healthy Subjects
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: No answer received from the Philippines Food and Drug Administration on protocol amendment issued due to IDMC recommendations. CYD vaccine 3rd dose not given.
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CYD66; U1111-1161-3294 (Other: WHO); 2019-003136-23 (EudraCT Number)
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Results first posted 2020-08-27 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Dengue Fever; Dengue Hemorrhagic Fever
Keywords: Dengue Fever; Dengue Hemorrhagic Fever; CYD Dengue Vaccine; Dengavaxia®
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — Dengue Vaccines; adacel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Concomitant Administration Group (Experimental): Participants will be administered the first dose of CYD dengue vaccine concomitantly with a dose of Tdap vaccine.
  Interventions: Biological: CYD Dengue Vaccine; Biological: Tdap: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine adsorbed
- Sequential Administration Group (Experimental): Participants will be administered the first dose of CYD dengue vaccine 28 days after a dose of Tdap vaccine.
  Interventions: Biological: CYD Dengue Vaccine; Biological: Tdap: Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed

INTERVENTIONS:
Biological: CYD Dengue Vaccine — 0.5 milliliter (mL), Subcutaneous at Month 1, 7 and Month 13, respectively
  Other Names: Dengvaxia®
Biological: Tdap: Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine adsorbed — 0.5 mL, intramuscularly (IM) at Month 1.
  Other Names: Adacel®
  Arms: Concomitant Administration Group
Biological: Tdap: Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed — 0.5 mL, intramuscularly at Day 0.
  Other Names: Adacel®
  Arms: Sequential Administration Group

SUMMARY:
The aim of the study was to investigate the immunogenicity and safety of CYD dengue vaccine and Tetanus Toxoid (T), Reduced Diphtheria Toxoid (D) and Acellular Pertussis Vaccine Adsorbed (ap) (Tdap) vaccine when both vaccines were administered concomitantly or sequentially.

Primary Objectives:

* To demonstrate the non-inferiority of the humoral immune response to the Tdap booster dose concomitantly administered with the first dose of CYD dengue vaccine as compared to sequential administration, measured 28 days after Tdap booster dose.
* To demonstrate the non-inferiority of the humoral immune response to the first dose of CYD dengue vaccine concomitantly administered with Tdap as compared to sequential administration, measured 28 days after the first dose of CYD dengue vaccine.

Secondary Objectives:

* To demonstrate the non-inferiority of the humoral immune response of 3 doses of CYD dengue vaccine with the first dose concomitantly administered with Tdap as compared to sequential administration, measured 28 days after the third dose of CYD dengue vaccine.
* To describe the humoral immune response at baseline and 28 days after the first and third doses of CYD dengue vaccine, in each and any group.
* To describe the humoral immune response of Tdap vaccine at baseline and 28 days after concomitant administration with the first dose of CYD dengue vaccine as compared to the sequential administration, in each and any group.
* To describe the safety of the CYD dengue vaccine and of the Tdap booster dose after each and any injection in each group.

DETAILED DESCRIPTION:
Participants were to receive CYD dengue vaccine according to a 3-dose schedule administered 6 months apart, with the first dose of CYD dengue vaccine administered either concomitantly or sequentially with a booster dose of the Tdap vaccine, Adacel®.

During the conduct of the study, a safety signal was identified which led to the Independent Data Monitoring Committee (IDMC) recommendation not to vaccinate participants who had never been infected by dengue prior to the first injection, i.e., dengue non-immune participants. The protocol was amended accordingly but never implemented due to absence of response of Health Authorities (HA) from The Philippines.

After having waited for more than 1.5 years, and as the participants became out of window to complete their immunization schedule and the last safety follow-up call (6 months after the last dose), the Sponsor decided to stop the trial. Participants only attended a last safety follow-up visit to terminate the study and were informed about the end of the study. As a consequence, the study was prematurely terminated before injection of the last dose (3rd dose) of the CYD dengue vaccine.

As a consequence of the IDMC recommendations, the main immunogenicity analyses were done in dengue immune participants which is not what was planned in the protocol (and this is why the primary endpoints are not exactly the same as those defined in the protocol as they were finally assessed only in dengue immune participants whereas initially it was planned to be assessed regardless of baseline status).

All participants were assessed for immunogenicity and safety. Safety assessments included solicited reactions within 7 or 14 days after each injection, unsolicited adverse events within 28 days after each injection, and serious adverse events during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged 9 to 60 years (i.e., from the day of the 9th birthday to the day prior to the 61th birthday) on the day of inclusion.
* Participant in good health, based on medical history and physical examination.
* Informed consent form (ICF) or assent form was signed and dated by the participant (based on local regulations), and/or ICF was signed and dated by the parent(s) or another legally acceptable representative (and by an independent witness if required by local regulations).
* For participant aged 9 to 11 years: known (documented) receipt of at least 4 previous doses of diphtheria toxoid, tetanus toxoid and acellular pertussis-containing (DTaP) vaccines, with the last dose not within the last 5 years prior to enrolment.

OR For participant aged at least 12 years: known (documented or self-reported) receipt of at least 3 previous doses of diphtheria toxoid, tetanus toxoid, and whole cell pertussis-containing (DTwP) vaccines, with the last dose not within the last 5 years prior to enrolment.

* Participant (or participant and parent[s]/legally acceptable representatives) was able to attend all scheduled visits and complied with all trial procedures.

Exclusion Criteria:

* Participant was pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination until at least 4 weeks after the last vaccination).
* Participation at the time of study enrollment (or in the 4 weeks preceding the first trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Planned receipt of any vaccine in the 4 weeks following any trial vaccination.
* Previous vaccination against dengue disease with the trial CYD dengue vaccine.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response.
* Known or suspected congenital or acquired immunodeficiency (including human immunodeficiency virus (HIV) infection with impaired immune function); or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroids therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* A previous severe reaction to pertussis, diphtheria or tetanus vaccine including immediate anaphylaxis, encephalopathy within 7 days or seizure within 3 days of receiving the vaccine.
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances.
* Thrombocytopenia, contraindicating IM vaccination.
* Bleeding disorder or receipt of anticoagulants within 3 weeks preceding inclusion, which might be a contraindication for IM vaccination, at the discretion of the Investigator.
* Deprived of freedom by administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction that, based on Investigator's judgment, may interfere with the participant's ability to comply with trial procedures.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with trial conduct or completion.
* Identified as an Investigator or employee of the Investigator with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.
* Self-reported HIV, Hepatitis B, or Hepatitis C infection.
* Personal history of Guillain-Barré syndrome.

Ages: 9 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 688 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (4):
- Philippines (4):
  - City of Muntinlupa, Alabang
  - Manila
  - Quezon
  - Quezon City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Santos J, Montellano ME, Solante R, Perreras N, Meyer S, Toh ML, Zocchetti C, Vigne C, Mascarenas C. Immunogenicity and Safety of a Tetravalent Dengue Vaccine Administered Concomitantly or Sequentially With Tdap Vaccine: Randomized Phase IIIb Trial in Healthy Participants 9-60 Years of Age in the Philippines. Pediatr Infect Dis J. 2021 Sep 1;40(9):856-863. doi: 10.1097/INF.0000000000003220. PMID 34117198

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 19 December 2016 to 17 April 2017 at 4 centers in the Philippines. A total of 688 participants were enrolled and randomized in this study.
Pre-assignment Details: Safety signal was spotted in dengue non-immune participants, which led to IDMC suggestion to not vaccinate them anymore. As no Health Authority feedback was received on amendment, study was terminated before 3rd (last) injection of CYD dengue vaccine. Hence, no participants received 3rd CYD dengue dose (as planned) and all were followed for safety.
Groups:
- CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration): Participants received 1 booster dose of Tetanus Toxoid (T), Reduced Diphtheria Toxoid (D) and Acellular Pertussis Vaccine Adsorbed (ap) (Tdap) vaccine 0.5 milliliter (mL) intramuscular (IM) injection at Month 1, and 2 doses of CYD dengue vaccine 0.5 mL subcutaneous (SC) injection at Month 1 (concomitantly with Tdap booster dose) and at Month 7.
- CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration): Participants received 1 booster dose of Tdap vaccine 0.5 mL IM injection at Day 0 and 2 doses of CYD dengue vaccine 0.5 mL SC injection at Month 1 (sequentially, one month after the Tdap booster dose) and at Month 7.
Period: Overall Study
Arm/Group | CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) | CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration)
Started | 346 | 342
Safety Analysis Set (SafAS) (SafAS: Participants who received at least one dose of the study vaccines (CYD and Tdap).) | 338 | 342
Completed | 0 | 0
Not Completed | 346 | 342
Not completed — Withdrawal by Subject | 11 | 12
Not completed — Non-compliance with the protocol | 308 | 308
Not completed — Lost to Follow-up | 27 | 22

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration): Participants received 1 booster dose of Tdap vaccine 0.5 mL IM injection at Month 1, and 2 doses of CYD dengue vaccine 0.5 mL SC injection at Month 1 (concomitantly with Tdap booster dose) and at Month 7.
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) | CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration) | Total
Number analyzed (Participants) | 346 | 342 | 688
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (16.3) | 27.1 (16.7) | 26.6 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187 | 193 | 380
  Male | 159 | 149 | 308
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Dengue Baseline Status [Count of Participants; unit: Participants] — Dengue immune participants were defined as participants with titers greater than or equal to (>=) 10 (1/dilution) for at least one serotype with the parental dengue virus strain. Dengue non-immune participants were defined as participants with titers less than (<) 10 (1/dilution) for all serotypes with parental dengue virus strains with available and 'valid' results.
  Participants
    Dengue immune | 314 | 315 | 629
    Dengue non-immune | 32 | 27 | 59

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentrations (GMCs) of Antibodies Against Pertussis Antigens (Pertussis Toxoid, Filamentous Hemagglutinin, Pertactin, and Fimbriae 2+3) 28 Days After Dose of Tdap Vaccine in Previously Dengue Immune Participants
Description: GMCs against each pertussis antigens (pertussis toxoid [PT], filamentous hemagglutinin [FHA], pertactin [PRN], fimbriae types 2 and 3 [FIM2+3]) were assessed using an enzyme-linked immunosorbent assay (ELISA) method and were measured in ELISA unit/milliliter (EU/mL). Dengue immune participants at Baseline were defined as participants with titers >=10 (1/dilution) for at least one serotype with the parental dengue virus strain.
Time Frame: 28 days after Tdap vaccination
Population: Per protocol analysis set of Tdap (PPT) included dengue immune participants who received at least one dose of Tdap and had no relevant protocol deviations. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) | CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration)
Number analyzed (Participants) | 312 | 314
EU/mL
  Anti-PT: number analyzed (Participants) | 300 | 310
  Anti-PT | 65.2 [57.7 to 73.8] | 76.0 [67.9 to 85.1]
  Anti-FHA: number analyzed (Participants) | 308 | 314
  Anti-FHA | 273 [248 to 299] | 267 [241 to 296]
  Anti-PRN: number analyzed (Participants) | 311 | 314
  Anti-PRN | 50.6 [41.4 to 61.9] | 44.9 [36.7 to 55.0]
  Anti-FIM2+3: number analyzed (Participants) | 309 | 312
  Anti-FIM2+3 | 705 [586 to 847] | 643 [537 to 770]
Statistical Analysis 1: Comparison: CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) vs CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration); Anti-PT; Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit of the two-sided 95% confidence interval (CI) of the ratio of GMCs between groups (Group 1/ Group 2) was greater than (>) 1/1.5 for each antigen. Overall non-inferiority was demonstrated if the 4 antigens achieved non-inferiority; GMC ratio = 0.848, 95% CI 2-sided [0.721 to 0.997]
Statistical Analysis 2: Comparison: CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) vs CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration); Anti-FHA; Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit of the two-sided 95% CI of the ratio of GMCs between groups (Group 1/ Group 2) was > 1/1.5 for each antigen. Overall non-inferiority was demonstrated if the 4 antigens achieved non-inferiority; GMC ratio = 1.02, 95% CI 2-sided [0.892 to 1.18]
Statistical Analysis 3: Comparison: CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) vs CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration); Anti-PRN; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMC ratio = 1.11, 95% CI 2-sided [0.836 to 1.46]
Statistical Analysis 4: Comparison: CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) vs CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration); Anti-FIM2+3; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMC ratio = 1.05, 95% CI 2-sided [0.827 to 1.33]

2. Primary Outcome: Percentage of Participants With Seroprotection Against Diphtheria and Tetanus Antigens 28 Days After the Dose of Tdap Vaccine in the Previously Dengue Immune Participants
Description: Seroprotection against diphtheria (Anti-D) and tetanus (Anti-T) antigens was performed by Micrometabolic Inhibition Test - Toxin Neutralization assay (MIT-TNA) and ELISA, respectively. Seroprotection was defined as anti-D and anti-T Ab concentration greater than 0.1 international units (IU)/mL. Dengue immune participants at Baseline were defined as participants with titers >=10 (1/dilution) for at least one serotype with the parental dengue virus strain.
Time Frame: 28 days after Tdap vaccination
Population: Analysis was performed on PPT population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) | CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration)
Number analyzed (Participants) | 312 | 314
percentage of participants
  Anti-D | 90.1 [86.2 to 93.1] | 89.8 [85.9 to 92.9]
  Anti-T: number analyzed (Participants) | 309 | 314
  Anti-T | 98.4 [96.3 to 99.5] | 99.0 [97.2 to 99.8]
Statistical Analysis 1: Comparison: CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) vs CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration); Anti-D; Test type: Non-Inferiority — The non-inferiority was demonstrated if the lower limit of all the 95% CI of the percentage difference was > -10% for all antigens; Percentage difference = 0.26, 95% CI 2-sided [-4.53 to 5.04]
Statistical Analysis 2: Comparison: CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) vs CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration); Anti-T; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage difference = -0.66, 95% CI 2-sided [-2.87 to 1.37]

3. Primary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Each Dengue Virus Serotype 28 Days After the First Dose of CYD Dengue Vaccination in the Previously Dengue Immune Participants
Description: The GMTs against each of the four parenteral dengue virus serotypes (1, 2, 3 and 4) of CYD dengue vaccine were assessed using the 50% plaque reduction neutralization test (PRNT50) assay method. Dengue immune participants at Baseline were defined as participants with titers >=10 (1/dilution) for at least one serotype with the parental dengue virus strain. Titers were measured in terms of 1/dilution.
Time Frame: 28 days after first CYD dengue vaccination
Population: Analysis was performed on per-protocol analysis set for CYD dengue vaccine (PPC) population which included dengue immune participants who received 1st dose of CYD dengue vaccine and had no relevant protocol deviations.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) | CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration)
Number analyzed (Participants) | 312 | 308
titers
  Serotype 1 | 513 [427 to 617] | 461 [384 to 552]
  Serotype 2 | 677 [588 to 780] | 568 [489 to 661]
  Serotype 3 | 653 [558 to 765] | 706 [603 to 828]
  Serotype 4 | 378 [324 to 442] | 472 [404 to 551]
Statistical Analysis 1: Comparison: CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) vs CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration); Serotype 1; Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit of the two-sided 95% CI of the ratio of GMTs between groups (Group 1/Group 2) was > 1/2 for each serotype. Overall non-inferiority was demonstrated if all 4 serotypes achieved non-inferiority; GMT ratio = 1.11, 95% CI 2-sided [0.862 to 1.44]
Statistical Analysis 2: Comparison: CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) vs CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration); Serotype 2; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.19, 95% CI 2-sided [0.97 to 1.47]
Statistical Analysis 3: Comparison: CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) vs CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration); Serotype 3; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; GMT ratio = 0.925, 95% CI 2-sided [0.739 to 1.16]
Statistical Analysis 4: Comparison: CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) vs CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration); Serotype 4; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; GMT ratio = 0.802, 95% CI 2-sided [0.644 to 0.999]

4. Secondary Outcome: Geometric Mean Titers of Antibodies Against Each Dengue Virus Serotype at Baseline and 28 Days After the First Dose of CYD Dengue Vaccination in the Previously Dengue Immune Participants
Description: The GMTs against each of the four parenteral dengue virus serotypes (1, 2, 3 and 4) of CYD dengue vaccine were assessed using PRNT50 assay method. Dengue immune participants at Baseline were defined as participants with titers >=10 (1/dilution) for at least one serotype with the parental dengue virus strain. Titers were measured in terms of 1/dilution.
Time Frame: Baseline (Pre-CYD vaccination 1) and 28 days after the first CYD dengue vaccination
Population: Analysis was performed on the subset of participants who received at least one dose of study vaccines (CYD dengue or Tdap) and were immune to dengue at baseline. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) | CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration)
Number analyzed (Participants) | 314 | 315
titers
  Serotype 1: Pre-vaccination 1 | 265 [218 to 322] | 250 [208 to 300]
  Serotype 1: 28 days post-vaccination 1: number analyzed (Participants) | 313 | 315
  Serotype 1: 28 days post-vaccination 1 | 513 [427 to 616] | 468 [392 to 560]
  Serotype 2: Pre-vaccination 1 | 404 [350 to 467] | 343 [294 to 401]
  Serotype 2: 28 days post-vaccination 1: number analyzed (Participants) | 313 | 315
  Serotype 2: 28 days post-vaccination 1 | 679 [589 to 781] | 577 [497 to 671]
  Serotype 3: Pre-vaccination 1 | 327 [274 to 391] | 327 [280 to 383]
  Serotype 3: 28 days post-vaccination 1: number analyzed (Participants) | 313 | 315
  Serotype 3: 28 days post-vaccination 1 | 655 [559 to 767] | 709 [605 to 830]
  Serotype 4: Pre-vaccination 1 | 136 [115 to 160] | 172 [150 to 197]
  Serotype 4: 28 days post-vaccination 1: number analyzed (Participants) | 313 | 315
  Serotype 4: 28 days post-vaccination 1 | 379 [325 to 443] | 478 [410 to 557]

5. Secondary Outcome: Percentage of Participants With Neutralizing Antibody Titers Against Each of the 4 Dengue Virus Serotypes of CYD at Baseline and 28 Days After First Dose of CYD Dengue Vaccination in the Previously Dengue Immune Participants
Description: The GMTs against each of the four parenteral dengue virus serotypes (1, 2, 3 and 4) of CYD dengue vaccine were assessed using PRNT50 assay method. Dengue immune participants at Baseline were defined as participants with titers >=10 (1/dilution) for at least one serotype with the parental dengue virus strain.
Time Frame: Baseline (Pre-CYD vaccination 1) and 28 days after the first CYD dengue vaccination
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) | CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration)
Number analyzed (Participants) | 314 | 315
percentage of participants
  Serotype 1: Pre-vaccination 1 | 92.7 [89.2 to 95.3] | 93.3 [90.0 to 95.8]
  Serotype 1: 28 days post-vaccination 1: number analyzed (Participants) | 313 | 315
  Serotype 1: 28 days post-vaccination 1 | 97.8 [95.4 to 99.1] | 98.4 [96.3 to 99.5]
  Serotype 2: Pre-vaccination 1 | 98.1 [95.9 to 99.3] | 96.5 [93.8 to 98.2]
  Serotype 2: 28 days post-vaccination 1: number analyzed (Participants) | 313 | 315
  Serotype 2: 28 days post-vaccination 1 | 100.0 [98.8 to 100.0] | 99.0 [97.2 to 99.8]
  Serotype 3: Pre-vaccination 1 | 95.5 [92.6 to 97.5] | 97.1 [94.6 to 98.7]
  Serotype 3: 28 days post-vaccination 1: number analyzed (Participants) | 313 | 315
  Serotype 3: 28 days post-vaccination 1 | 100.0 [98.8 to 100.0] | 99.7 [98.2 to 100.0]
  Serotype 4: Pre-vaccination 1 | 93.0 [89.6 to 95.6] | 97.5 [95.1 to 98.9]
  Serotype 4: 28 days post-vaccination 1: number analyzed (Participants) | 313 | 315
  Serotype 4: 28 days post-vaccination 1 | 99.4 [97.7 to 99.9] | 100.0 [98.8 to 100.0]

6. Secondary Outcome: Percentage of Participants With Neutralizing Antibody Titers Above Predefined Thresholds Against at Least 1, 2, 3, or 4 Serotypes of CYD at Baseline and 28 Days After the First Dose of CYD Dengue Vaccination in the Previously Dengue Immune Participants
Description: Dengue neutralizing antibody levels against each of the 4 dengue virus serotypes (1, 2, 3, and 4) were measured by PRNT50. Dengue immune participants at Baseline were defined as participants with titers >=10 (1/dilution) for at least one serotype with the parental dengue virus strain. Percentage of participants with neutralizing antibody titers above pre-defined thresholds (>=10 and >=100 [1/dilution]) against at least 1, 2, 3, or 4 serotypes of CYD were reported. Here, 'dil'=dilution and "vac"=vaccination in the specified categories.
Time Frame: Baseline (Pre-CYD vaccination 1) and 28 days after the first CYD dengue vaccination
Population: Analysis was performed on subset of participants who received at least one dose of study vaccines (CYD dengue or Tdap) and were immune to dengue at baseline. Here, 'Number analyzed' = participants with available data for each specified categories.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) | CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration)
Number analyzed (Participants) | 314 | 315
percentage of participants
  At least 1 Serotype: pre-vac 1: >=10 (1/dil) | 100.0 [98.8 to 100.0] | 100.0 [98.8 to 100.0]
  At least 1 Serotype: pre-vac1: >=100 (1/dil) | 97.8 [95.5 to 99.1] | 97.1 [94.6 to 98.7]
  At least 1 Serotype: post-vac 1: >=10 (1/dil): number analyzed (Participants) | 313 | 315
  At least 1 Serotype: post-vac 1: >=10 (1/dil) | 100.0 [98.8 to 100.0] | 100.0 [98.8 to 100.0]
  At least 1 Serotype: post-vac 1: >=100 (1/dil): number analyzed (Participants) | 313 | 315
  At least 1 Serotype: post-vac 1: >=100 (1/dil) | 99.7 [98.2 to 100.0] | 99.7 [98.2 to 100.0]
  At least 2 Serotype: pre-vac 1: >=10 (1/dil) | 96.5 [93.8 to 98.2] | 98.1 [95.9 to 99.3]
  At least 2 Serotype: pre-vac 1: >=100 (1/dil) | 84.4 [79.9 to 88.2] | 87.0 [82.8 to 90.5]
  At least 2 Serotype: post-vac 1: >=10 (1/dil): number analyzed (Participants) | 313 | 315
  At least 2 Serotype: post-vac 1: >=10 (1/dil) | 100.0 [98.8 to 100.0] | 99.7 [98.2 to 100.0]
  At least 2 Serotype: post-vac 1: >=100 (1/dil): number analyzed (Participants) | 313 | 315
  At least 2 Serotype: post-vac 1: >=100 (1/dil) | 95.8 [93.0 to 97.8] | 96.5 [93.8 to 98.2]
  At least 3 Serotype: pre-vac 1: >=10 (1/dil) | 93.6 [90.3 to 96.1] | 95.2 [92.3 to 97.3]
  At least 3 Serotype: pre-vac 1: >=100 (1/dil) | 76.1 [71.0 to 80.7] | 76.8 [71.8 to 81.4]
  At least 3 Serotype: post-vac 1: >=10 (1/dil): number analyzed (Participants) | 313 | 315
  At least 3 Serotype: post-vac 1: >=10 (1/dil) | 99.7 [98.2 to 100.0] | 99.4 [97.7 to 99.9]
  At least 3 Serotype: post-vac 1: >=100 (1/dil): number analyzed (Participants) | 313 | 315
  At least 3 Serotype: post-vac 1: >=100 (1/dil) | 90.4 [86.6 to 93.4] | 92.1 [88.5 to 94.8]
  At least 4 Serotype: pre-vac 1: >=10 (1/dil) | 89.2 [85.2 to 92.4] | 91.1 [87.4 to 94.0]
  At least 4 Serotype: pre-vac 1: >=100 (1/dil) | 52.9 [47.2 to 58.5] | 54.3 [48.6 to 59.9]
  At least 4 Serotype: post-vac 1: >=10 (1/dil): number analyzed (Participants) | 313 | 315
  At least 4 Serotype: post-vac 1: >=10 (1/dil) | 97.4 [95.0 to 98.9] | 98.1 [95.9 to 99.3]
  At least 4 Serotype: post-vac 1: >=100 (1/dil): number analyzed (Participants) | 313 | 315
  At least 4 Serotype: post-vac 1: >=100 (1/dil) | 73.8 [68.6 to 78.6] | 75.6 [70.4 to 80.2]

7. Secondary Outcome: Geometric Mean Concentrations of Serum Antibodies Against Pertussis Antigens (Pertussis Toxoid, Filamentous Hemagglutinin, Pertactin, and Fimbriae 2+3) at Baseline and 28 Days After the Dose of Tdap Vaccine in the Previously Dengue Immune Participants
Description: GMCs against each pertussis antigens (PT, FHA, PRN, FIM2+3) were assessed using ELISA assay method and were measured in EU/mL. Dengue immune participants at Baseline were defined as participants with titers >=10 (1/dilution) for at least one serotype with the parental dengue virus strain.
Time Frame: Baseline (Pre-Tdap vaccination) and 28 days after the Tdap vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) | CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration)
Number analyzed (Participants) | 314 | 315
EU/mL
  Anti-PT: Pre-vaccination: number analyzed (Participants) | 313 | 313
  Anti-PT: Pre-vaccination | 8.46 [7.34 to 9.75] | 9.56 [8.33 to 11.0]
  Anti-PT: 28 days post-vaccination: number analyzed (Participants) | 301 | 311
  Anti-PT: 28 days post-vaccination | 65.0 [57.5 to 73.5] | 76.1 [68.1 to 85.2]
  Anti-FHA: Pre-vaccination: number analyzed (Participants) | 310 | 314
  Anti-FHA: Pre-vaccination | 19.9 [17.6 to 22.6] | 19.4 [17.1 to 22.1]
  Anti-FHA: 28 days post-vaccination: number analyzed (Participants) | 309 | 315
  Anti-FHA: 28 days post-vaccination | 272 [248 to 299] | 266 [240 to 295]
  Anti-PRN: Pre-vaccination | 3.79 [3.39 to 4.24] | 3.65 [3.25 to 4.10]
  Anti-PRN: 28 days post-vaccination: number analyzed (Participants) | 312 | 315
  Anti-PRN: 28 days post-vaccination | 50.6 [41.4 to 61.8] | 45.0 [36.8 to 55.1]
  Anti-FIM2+3: Pre-vaccination: number analyzed (Participants) | 297 | 298
  Anti-FIM2+3: Pre-vaccination | 15.1 [12.4 to 18.5] | 14.9 [12.2 to 18.1]
  Anti-FIM2+3: 28 days post-vaccination: number analyzed (Participants) | 310 | 313
  Anti-FIM2+3: 28 days post-vaccination | 700 [583 to 841] | 642 [537 to 769]

8. Secondary Outcome: Percentage of Participants Achieving Serum Antibody (>=0.1 IU/mL) Against Diphtheria and Tetanus Antigens at Baseline and 28 Days After the Dose of Tdap Vaccine in the Previously Dengue Immune Participants
Description: The GMC against diphtheria and tetanus antigens was performed by MIT-TNA and ELISA, respectively. Dengue immune participants at Baseline were defined as participants with titers >=10 (1/dilution) for at least one serotype with the parental dengue virus strain.
Time Frame: Baseline (Pre-Tdap vaccination) and 28 days after the dose of Tdap vaccination
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) | CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration)
Number analyzed (Participants) | 314 | 315
percentage of participants
  Anti-D: Pre-vaccination: number analyzed (Participants) | 314 | 314
  Anti-D: Pre-vaccination | 31.8 [26.7 to 37.3] | 32.8 [27.6 to 38.3]
  Anti-T: Pre-vaccination: number analyzed (Participants) | 314 | 313
  Anti-T: Pre-vaccination | 63.7 [58.1 to 69.0] | 69.6 [64.2 to 74.7]
  Anti-D: 28 days post-vaccination: number analyzed (Participants) | 313 | 315
  Anti-D: 28 days post-vaccination | 90.1 [86.2 to 93.2] | 89.8 [86.0 to 92.9]
  Anti-T: 28 days post-vaccination: number analyzed (Participants) | 310 | 315
  Anti-T: 28 days post-vaccination | 98.1 [95.8 to 99.3] | 99.0 [97.2 to 99.8]

9. Secondary Outcome: Number of Participants With Immediate Unsolicited Adverse Events (AE) Following Vaccination With Tdap or CYD Dengue Vaccine
Description: An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the electronic case report form (eCRF) in terms of diagnosis and/or onset post-vaccination. Any unsolicited AE occurred during first 30 minutes post-vaccination was recorded on the CRF as immediate AE. At Visit 1, participants of Group 1 received no vaccination and participants of Group 2 received only Tdap vaccination. At Visit 2, participants of Group 1 received both CYD and Tdap vaccination and participants of Group 2 received only CYD vaccination. At Visit 4, participants of Groups 1 and 2 received CYD vaccination.
Time Frame: Within 30 minutes after any and each vaccination
Population: Analysis was performed on SafAS population, which included participants who received at least one dose of the study vaccines (CYD dengue or Tdap). Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) | CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration)
Number analyzed (Participants) | 338 | 342
Participants
  Post any vaccination | 0 | 0
  Post Tdap vaccination 1 (Visit 1): number analyzed (Participants) | 0 | 342
  Post Tdap vaccination 1 (Visit 1) |  | 0
  Post CYD/Tdap vaccination (Visit 2): number analyzed (Participants) | 338 | 338
  Post CYD/Tdap vaccination (Visit 2) | 0 | 0
  Post CYD vaccination 2 (Visit 4): number analyzed (Participants) | 321 | 319
  Post CYD vaccination 2 (Visit 4) | 0 | 0

10. Secondary Outcome: Number of Participants With Solicited Injection Site Reactions Following Vaccination With Tdap or CYD Dengue Vaccine
Description: A solicited reaction (SR) was an AE observed and reported under the conditions (symptom and onset) prelisted (i.e., solicited) in the eCRF and considered as related to vaccination. Solicited injection site reactions included pain, erythema, and swelling. At Visit 1, participants of Group 1 received no vaccination and participants of Group 2 received only Tdap vaccination. At Visit 2, participants of Group 1 received both CYD and Tdap vaccinations and participants of Group 2 received only CYD vaccination. At Visit 4, participants of Groups 1 and 2 received only CYD vaccination.
Time Frame: Within 7 days after any and each vaccination
Population: Analysis was performed on SafAS population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) | CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration)
Number analyzed (Participants) | 338 | 342
Participants
  Pain: Post any vaccination: number analyzed (Participants) | 338 | 341
  Pain: Post any vaccination | 229 | 237
  Pain: Post Tdap vaccination (Visit 1): number analyzed (Participants) | 0 | 341
  Pain: Post Tdap vaccination (Visit 1) |  | 212
  Pain: Post CYD/Tdap vaccination (Visit 2): number analyzed (Participants) | 338 | 338
  Pain: Post CYD/Tdap vaccination (Visit 2) | 218 | 53
  Pain: Post CYD vaccination 2 (Visit 4): number analyzed (Participants) | 320 | 319
  Pain: Post CYD vaccination 2 (Visit 4) | 61 | 55
  Erythema: Post any vaccination: number analyzed (Participants) | 338 | 341
  Erythema: Post any vaccination | 14 | 17
  Erythema: Post Tdap vaccination (Visit 1): number analyzed (Participants) | 0 | 341
  Erythema: Post Tdap vaccination (Visit 1) |  | 14
  Erythema: Post CYD/Tdap vaccination (Visit 2): number analyzed (Participants) | 338 | 338
  Erythema: Post CYD/Tdap vaccination (Visit 2) | 13 | 5
  Erythema: Post CYD vaccination 2 (Visit 4): number analyzed (Participants) | 320 | 319
  Erythema: Post CYD vaccination 2 (Visit 4) | 2 | 2
  Swelling: Post any vaccination: number analyzed (Participants) | 338 | 341
  Swelling: Post any vaccination | 25 | 32
  Swelling: Post Tdap vaccination (Visit 1): number analyzed (Participants) | 0 | 341
  Swelling: Post Tdap vaccination (Visit 1) |  | 30
  Swelling: Post CYD/Tdap vaccination (Visit 2): number analyzed (Participants) | 338 | 338
  Swelling: Post CYD/Tdap vaccination (Visit 2) | 25 | 3
  Swelling: Post CYD vaccination 2 (Visit 4): number analyzed (Participants) | 320 | 319
  Swelling: Post CYD vaccination 2 (Visit 4) | 2 | 2

11. Secondary Outcome: Number of Participants With Solicited Systemic Reactions Following Vaccination With Tdap or CYD Dengue Vaccine
Description: A SR reaction was an AE observed and reported under the conditions (symptom and onset) prelisted (i.e., solicited) in the CRF and considered as related to vaccination. Solicited injection site reactions included fever, headache, malaise, myalgia, and asthenia. At Visit 1, participants of Group 1 received no vaccination and participants of Group 2 received only Tdap vaccination. At Visit 2, participants of Group 1 received both CYD and Tdap vaccinations and participants of Group 2 received only CYD vaccination. At Visit 4, participants of Groups 1 and 2 received only CYD vaccination.
Time Frame: Within 14 days after any and each vaccination
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) | CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration)
Number analyzed (Participants) | 338 | 342
Participants
  Fever: Post any vaccination: number analyzed (Participants) | 338 | 340
  Fever: Post any vaccination | 21 | 30
  Fever: Post Tdap vaccination (Visit 1): number analyzed (Participants) | 0 | 339
  Fever: Post Tdap vaccination (Visit 1) |  | 15
  Fever: Post CYD/Tdap vaccination (Visit 2): number analyzed (Participants) | 338 | 338
  Fever: Post CYD/Tdap vaccination (Visit 2) | 11 | 6
  Fever: Post CYD vaccination 2 (Visit 4): number analyzed (Participants) | 320 | 319
  Fever: Post CYD vaccination 2 (Visit 4) | 10 | 9
  Headache: Post any vaccination: number analyzed (Participants) | 338 | 341
  Headache: Post any vaccination | 89 | 115
  Headache: Post Tdap vaccination (Visit 1): number analyzed (Participants) | 0 | 341
  Headache: Post Tdap vaccination (Visit 1) |  | 83
  Headache: Post CYD/Tdap vaccination (Visit 2): number analyzed (Participants) | 338 | 338
  Headache: Post CYD/Tdap vaccination (Visit 2) | 70 | 33
  Headache: Post CYD vaccination 2 (Visit 4): number analyzed (Participants) | 320 | 319
  Headache: Post CYD vaccination 2 (Visit 4) | 36 | 35
  Malaise: Post any vaccination: number analyzed (Participants) | 338 | 341
  Malaise: Post any vaccination | 91 | 111
  Malaise: Post Tdap vaccination (Visit 1): number analyzed (Participants) | 0 | 341
  Malaise: Post Tdap vaccination (Visit 1) |  | 81
  Malaise: Post CYD/Tdap vaccination (Visit 2): number analyzed (Participants) | 338 | 338
  Malaise: Post CYD/Tdap vaccination (Visit 2) | 74 | 28
  Malaise: Post CYD vaccination 2 (Visit 4): number analyzed (Participants) | 320 | 319
  Malaise: Post CYD vaccination 2 (Visit 4) | 32 | 33
  Myalgia: Post any vaccination: number analyzed (Participants) | 338 | 341
  Myalgia: Post any vaccination | 74 | 100
  Myalgia: Post Tdap vaccination (Visit 1): number analyzed (Participants) | 0 | 341
  Myalgia: Post Tdap vaccination (Visit 1) |  | 78
  Myalgia: Post CYD/Tdap vaccination (Visit 2): number analyzed (Participants) | 338 | 338
  Myalgia: Post CYD/Tdap vaccination (Visit 2) | 67 | 30
  Myalgia: Post CYD vaccination 2 (Visit 4): number analyzed (Participants) | 320 | 319
  Myalgia: Post CYD vaccination 2 (Visit 4) | 26 | 22
  Asthenia: Post any vaccination: number analyzed (Participants) | 338 | 341
  Asthenia: Post any vaccination | 67 | 94
  Asthenia: Post Tdap vaccination (Visit 1): number analyzed (Participants) | 0 | 341
  Asthenia: Post Tdap vaccination (Visit 1) |  | 69
  Asthenia: Post CYD/Tdap vaccination (Visit 2): number analyzed (Participants) | 338 | 338
  Asthenia: Post CYD/Tdap vaccination (Visit 2) | 59 | 24
  Asthenia: Post CYD vaccination 2 (Visit 4): number analyzed (Participants) | 320 | 319
  Asthenia: Post CYD vaccination 2 (Visit 4) | 19 | 22

12. Secondary Outcome: Number of Participants Reporting Unsolicited Adverse Events Following Vaccination With Tdap or CYD Dengue Vaccine
Description: An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the eCRF in terms of diagnosis and/or onset post-vaccination. At Visit 1, participants of Group 1 received no vaccination and participants of Group 2 received only Tdap vaccination. At Visit 2, participants of Group 1 received both CYD and Tdap vaccinations and participants of Group 2 received only CYD vaccination. At Visit 4, participants of Groups 1 and 2 received CYD vaccination.
Time Frame: Within 28 days after any and each vaccination
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) | CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration)
Number analyzed (Participants) | 338 | 342
Participants
  Post any vaccination | 56 | 70
  Post Tdap vaccination (Visit 1): number analyzed (Participants) | 0 | 342
  Post Tdap vaccination (Visit 1) |  | 40
  Post CYD/Tdap vaccination (Visit 2): number analyzed (Participants) | 338 | 338
  Post CYD/Tdap vaccination (Visit 2) | 37 | 20
  Post CYD vaccination 2 (Visit 4): number analyzed (Participants) | 321 | 319
  Post CYD vaccination 2 (Visit 4) | 28 | 26

13. Secondary Outcome: Number of Participants Reporting Non-serious Adverse Event of Special Interests (AESIs) Following Vaccination With Tdap or CYD Dengue Vaccine
Description: Non-serious AESIs were non-serious AEs that were considered by the Sponsor to be relevant for the monitoring of the safety profile of the investigational vaccine. At Visit 1, participants of Group 1 received no vaccination and participants of Group 2 received only Tdap vaccination. At Visit 2, participants of Group 1 received both CYD and Tdap vaccinations and participants of Group 2 received only CYD vaccination. At Visit 4, participants of Groups 1 and 2 received CYD vaccination.
Time Frame: Within 7 days post any and each vaccination
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) | CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration)
Number analyzed (Participants) | 338 | 342
Participants
  Post any vaccination | 0 | 0
  Post Tdap vaccination (Visit 1): number analyzed (Participants) | 0 | 342
  Post Tdap vaccination (Visit 1) |  | 0
  Post CYD/Tdap vaccination (Visit 2): number analyzed (Participants) | 338 | 338
  Post CYD/Tdap vaccination (Visit 2) | 0 | 0
  Post CYD vaccination 2 (Visit 4): number analyzed (Participants) | 321 | 319
  Post CYD vaccination 2 (Visit 4) | 0 | 0

14. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs) and Serious AESIs Following Vaccination With Tdap or CYD Dengue Vaccine
Description: SAEs were AEs resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening; required hospitalization or prolonged existing hospitalization; persistent or significant disability/incapacity; congenital anomaly or a medically important event. Serious AESIs were SAEs that were considered by the Sponsor to be relevant for the monitoring of the safety profile of the investigational vaccine.
Time Frame: From Day 0 up to 6 months after the last Tdap or CYD vaccination
Population: Analysis was performed on SafAS population.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) | CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration)
Number analyzed (Participants) | 338 | 342
Participants
  SAE | 8 | 11
  Serious AESI | 1 | 3

15. Secondary Outcome: Number of Participants Reporting Cases of Virologically Confirmed Dengue (VCD) Hospitalization Following Vaccination With Tdap or CYD Dengue Vaccine
Description: Hospitalized suspected dengue case was defined as an acute febrile illness with diagnosis of dengue requiring hospitalization (with bed attribution). In such cases, 1 unplanned acute blood sample (within the first 5 days after fever onset) was collected for virological confirmation of hospitalized suspected dengue case. A suspected case was considered VCD if there was a detection of wild type dengue virus by dengue non-structural protein 1 antigen ELISA and/or dengue reverse transcriptase-polymerase chain reactions.
Time Frame: From Day 0 up to 6 months after the last Tdap or CYD vaccination
Population: Analysis was performed on SafAS population.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) | CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration)
Number analyzed (Participants) | 338 | 342
Participants | 0 | 3

ADVERSE EVENTS:
Time Frame: AE data were collected from Day 0 up to Day 28 post any vaccination. SR data were collected from Day 0 up to Day 14 post-vaccination. The SAEs were collected throughout the trial, i.e. up to 6 months after last Tdap or CYD vaccination.
Description: SR was an AE that was prelisted (i.e., solicited) in the eCRF and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the CRF (i.e., solicited) in terms of symptom and/or onset post-vaccination. Analysis was performed on SafAS population.
Arm/Group | CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) | CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration)
All-Cause Mortality (participants affected / at risk) | 0/338 | 0/342
Serious Adverse Events (participants affected / at risk) | 8/338 | 11/342
Other Adverse Events (participants affected / at risk) | 248/338 | 263/342
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) (N=338) | CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration) (N=342)
Hypertensive Heart Disease (Cardiac disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Jaundice Cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Atypical Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Dengue Fever (Infections and infestations) | 1 (1) | 3 (3)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Incisional Hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Abortion Complete (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Rash Generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine + Tdap Vaccine (Concomitant Administration) (N=338) | CYD Dengue Vaccine + Tdap Vaccine (Sequential Administration) (N=342)
Asthenia (General disorders) | 67 (78) | 94 (115)
Injection Site Pain (General disorders) | 229 (376) | 237 (320)
Injection Site Swelling (General disorders) | 25 (29) | 32 (35)
Malaise (General disorders) | 91 (106) | 111 (142)
Pyrexia (General disorders) | 22 (22) | 32 (33) — Pyrexia/fever events that occurred after 14 days post-vaccination were considered as unsolicited AEs.
Upper Respiratory Tract Infection (Infections and infestations) | 17 (17) | 17 (21)
Myalgia (Musculoskeletal and connective tissue disorders) | 74 (93) | 100 (130)
Headache (Nervous system disorders) | 89 (106) | 116 (152) — Headache event that occurred after 14 days post-vaccination was considered as an unsolicited AE.

LIMITATIONS AND CAVEATS:
Due to absence of response of competent authorities from The Philippines on protocol amendment, the study was prematurely terminated before injection of last dose (3rd dose) of the CYD dengue vaccine. Objectives related to 3rd dose were not assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/18/NCT02992418/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT02992418/SAP_001.pdf